CLINICAL TRIAL: NCT03130764
Title: Identification of Tumor Neoantigens During Immune Checkpoint Blockade in Resectable Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Durvalumab and Tremelimumab for Adjuvant Therapy of Resected NSCLC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI Transferred
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAQ8535
Record Dates: First submitted 2017-04-04; First posted 2017-04-26 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Durvalumab/Tremelimumab (Experimental): Patients with resected stage IB-IIIA NSCLC who have completed standard adjuvant therapy (as recommended by the treating physician) to receive durvalumab-tremelimumab will be enrolled. Patients will receive durvalumab (20 mg/kg) intravenously every 4 weeks for 1 year and tremelimumab (1 mg/kg) intravenously every 4 weeks for 4 doses.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Drug: Durvalumab — 1500 mg, IV over 1 hour Every 4 weeks for 1 year
  Other Names: MEDI4736
Drug: Tremelimumab — 75 mg, IV over 1 hour Every 4 weeks for 4 doses
  Other Names: CP-675,206

SUMMARY:
Despite aggressive surgery and chemotherapy, the risk of lung cancer recurrence remains high in most patients. This study aims to determine if a novel immune therapy consisting of two drugs is feasible and potentially increases the chance of cure in lung cancer patients after surgery and standard chemotherapy. The immune-based therapy being given in this study consists of two medications named durvalumab and tremelimumab.

DETAILED DESCRIPTION:
Lung cancer is the most common cancer and leading cause of cancer related death worldwide, accounting for more than 1.3 million deaths annually. The 5 year survival of clinical stage IIIA NSCLC, a technically curable lung cancer by surgery, chemotherapy +/- radiotherapy delivered in the perioperative setting, remains a modest 15%, with systemic recurrence occurring in the majority of patients. 5 year overall survival (OS) for patients with stage IB and II disease is also modest at 53% and 25% respectively.

The FDA approvals of T-cell checkpoint inhibitors, targeting programmed cell death-1 (PD-1) has changed the landscape of NSCLC. Although robust responses to anti-PD-1 can be observed, it is a small subset of patients with durable benefit. In phase 3 trials, the response rate to anti-PD- 1 is 19% with only ½ of these patients experiencing durable benefit. Even NSCLC tumors with high levels of PD-L1 have only a 30% response rate and combination immunotherapy has improved efficacy modestly.

Clinical trials in resectable lung cancer, have traditionally attempted to institute new agents in the adjuvant setting. However clinical endpoints take years of follow-up to ascertain. For example, The ANITA study was the most recent phase III study of adjuvant chemotherapy in NSCLC. In this study, results were published 12 years after study initiation. Thus, while OS remains the gold standard for assessment of benefit of adjuvant therapy, studies that are 12 years long are slow, expensive, and may yield results that are out of date by the time they are published. Thus the use of valid surrogate endpoints for OS is a high priority in NSCLC.

The potential for durable benefit in the advanced NSCLC setting has, not unexpectably, led to a foray with immune checkpoint blockade treatment into the adjuvant setting for resectable NSCLC. Randomized trials with durvalumab, pembrolizumab, and nivolumab are all underway.

However in the resected setting, adjuvant patients cannot be monitored radiologically for treatment response due to the absence of measurable disease thus requiring innovative in vitro and in vivo methods to study therapeutic response to immune checkpoint blockade. Encouragingly, as proof of concept, single-agent ipilimumab has demonstrated improved recurrence-free survival at 3 years in resected stage III melanoma compared to placebo leading to FDA approval in this setting. Less encouragingly, the hazard ratio favored the higher risk patients suggesting the benefit may be restricted to those tumors more apt to have residual disease and may represent the subset where benefit is most realized. Furthermore the data are not sufficiently mature to demonstrate an overall survival advantage nor is it known if this data can be extrapolated to NSCLC where responses are numerically lower.

Patients with resectable NSCLC will undergo surgical resection and bone marrow procurement at the same time. Tumor will be dissociated into single cell suspension and separated into viable cryopreserved tumor cells and tumor infiltrating lymphocytes will be expanded in media and high dose IL-2. Post-operatively, after recovery from surgical resection, patients will receive adjuvant treatment with chemotherapy as determined by the treating physician. Subsequently patients will receive adjuvant durvalumab for 12 doses and tremelimumab for 4 doses. Serial PBMCs will be obtained every 4 weeks during therapy. Primary resected tumor will undergo whole exome sequencing and RNA sequencing and clonal neoantigens will be predicted with established algorithms. Neoantigen specific T cell reactivity will be tested in autologous PBMCs with multimer (quantitative) and ICS (functional) assays.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and any locally-required authorization (e.g., HIPAA in the USA, EU Data Privacy Directive in the EU) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
* Adequate tissue must have been obtained from surgical intervention to satisfy biospecimen requirements of study (collected under biospecimen collection protocols; either AAAO5706 or AAAR1327).
* Histologically or cytologically confirmed squamous or non-squamous NSCLC.
* Stage IB-IIIA
* R0 or R1 resection
* Patients must have completed surgical resection and adjuvant chemotherapy (adjuvant radiotherapy excluded) with no significant persisting treatment related toxicity (grade 1 toxicity per CTCAE v4.0 allowed) as determined by the treating physician.
* Study treatment must begin within 30 days of surgical resection or adjuvant treatment. This timeline may be extended if further time for recovery from treatment related toxicities is required.
* Age ≥18 years; as no dosing or adverse event data are currently available on the use of durvalumab-tremelimumab in patients <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* ECOG performance status ≤1 (Karnofsky ≥70%).
* Patients must have normal organ and marrow function as defined below:

  * Hemoglobin >or = 9.0 g/dL
  * Absolute neutrophil count ≥1.5 x 109/L
  * Platelets ≥100 x 109/L
  * Total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * Serum creatinine CL > or = 40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance.
* The effects of durvalumab-tremelimumab on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and 6 months after completion of durvalumab + tremelimumab administration or 90 days after the last dose of durvalumab monotherapy, whichever is the longer time period. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of durvalumab + tremelimumab administration or 90 days after the last dose of durvalumab monotherapy, whichever is the longer time period.
* Ability to understand and the willingness to sign a written informed consent document.
* Female subjects must either be of non-reproductive potential (ie, post-menopausal by history: ≥60 years old and no menses for ≥1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

* Pre- or post-operative radiotherapy.
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
* Participation in another clinical study with an investigational product during the last 4 weeks
* Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab or an anti-CTLA4, including tremelimumab
* Mean QT interval corrected for heart rate (QTc) ≥ 470 ms calculated from 3 electrocardiograms (ECGs) using Fredericia's Correction
* Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab or tremelimumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
* Any unresolved toxicity ( > CTCAE grade 2) from previous anti-cancer therapy.
* Any prior Grade ≥ 3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1
* Active or prior documented autoimmune disease within the past 2 years NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
* Active hepatitis B or C (defined as positive Hepatitis B surface antigen, hepatitis C antibody)
* History of HIV infection
* History of interstitial lung disease/pneumonitis from any cause
* Never-smokers if EGFR/ALK testing results are unknown
* Patients with NSCLC that harbors an ALK rearrangement, or sensitizing EGFR mutation.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because durvalumab-tremelimumab are investigational agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with durvalumab-tremelimumab, breastfeeding should be discontinued if the mother is treated with these agents.
* History of allogeneic organ transplant
* History of hypersensitivity to durvalumab or any excipient
* History of hypersensitivity to the combination or comparator agent
* Known history of active tuberculosis
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab or tremelimumab
* Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of durvalumab + tremelimumab combination therapy or 90 days after the last dose of durvalumab monotherapy, whichever is the longer time period

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03 (Estimated); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
The percentage rate of induced T-cell response in resected NSCLC patients | Upto 1 year
  An induced T-cell response is defined as T-cell activity against a tumor neoantigen detected in T-cells isolated from PBMCs collected at any timepoint after initiation of durvalumab-tremelimumab.

SECONDARY OUTCOMES:
Percentage of patients that complete at least 80% of the prescribed study treatments. | Upto 2 years
  Feasibility of adjuvant therapy with druvalumab-tremelimumab
Disease Free Survival Rate (DFS) | Upto 12 Months
  Defined as the time from randomization until either disease recurrence at any site or death.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Sacher, M.D., Principal Investigator — Columbia University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Antonia S, Goldberg SB, Balmanoukian A, Chaft JE, Sanborn RE, Gupta A, Narwal R, Steele K, Gu Y, Karakunnel JJ, Rizvi NA. Safety and antitumour activity of durvalumab plus tremelimumab in non-small cell lung cancer: a multicentre, phase 1b study. Lancet Oncol. 2016 Mar;17(3):299-308. doi: 10.1016/S1470-2045(15)00544-6. Epub 2016 Feb 6. PMID 26858122
- [Background] Ferlay J, Shin HR, Bray F, Forman D, Mathers C, Parkin DM. Estimates of worldwide burden of cancer in 2008: GLOBOCAN 2008. Int J Cancer. 2010 Dec 15;127(12):2893-917. doi: 10.1002/ijc.25516. PMID 21351269
- [Background] Goldstraw P, Crowley J, Chansky K, Giroux DJ, Groome PA, Rami-Porta R, Postmus PE, Rusch V, Sobin L; International Association for the Study of Lung Cancer International Staging Committee; Participating Institutions. The IASLC Lung Cancer Staging Project: proposals for the revision of the TNM stage groupings in the forthcoming (seventh) edition of the TNM Classification of malignant tumours. J Thorac Oncol. 2007 Aug;2(8):706-14. doi: 10.1097/JTO.0b013e31812f3c1a. PMID 17762336
- [Background] Borghaei H, Paz-Ares L, Horn L, Spigel DR, Steins M, Ready NE, Chow LQ, Vokes EE, Felip E, Holgado E, Barlesi F, Kohlhaufl M, Arrieta O, Burgio MA, Fayette J, Lena H, Poddubskaya E, Gerber DE, Gettinger SN, Rudin CM, Rizvi N, Crino L, Blumenschein GR Jr, Antonia SJ, Dorange C, Harbison CT, Graf Finckenstein F, Brahmer JR. Nivolumab versus Docetaxel in Advanced Nonsquamous Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Oct 22;373(17):1627-39. doi: 10.1056/NEJMoa1507643. Epub 2015 Sep 27. PMID 26412456
- [Background] Herbst RS, Baas P, Kim DW, Felip E, Perez-Gracia JL, Han JY, Molina J, Kim JH, Arvis CD, Ahn MJ, Majem M, Fidler MJ, de Castro G Jr, Garrido M, Lubiniecki GM, Shentu Y, Im E, Dolled-Filhart M, Garon EB. Pembrolizumab versus docetaxel for previously treated, PD-L1-positive, advanced non-small-cell lung cancer (KEYNOTE-010): a randomised controlled trial. Lancet. 2016 Apr 9;387(10027):1540-1550. doi: 10.1016/S0140-6736(15)01281-7. Epub 2015 Dec 19. PMID 26712084
- [Background] Eggermont AM, Chiarion-Sileni V, Grob JJ, Dummer R, Wolchok JD, Schmidt H, Hamid O, Robert C, Ascierto PA, Richards JM, Lebbe C, Ferraresi V, Smylie M, Weber JS, Maio M, Konto C, Hoos A, de Pril V, Gurunath RK, de Schaetzen G, Suciu S, Testori A. Adjuvant ipilimumab versus placebo after complete resection of high-risk stage III melanoma (EORTC 18071): a randomised, double-blind, phase 3 trial. Lancet Oncol. 2015 May;16(5):522-30. doi: 10.1016/S1470-2045(15)70122-1. Epub 2015 Mar 31. PMID 25840693